CLINICAL TRIAL: NCT05909644
Title: A Single Sequence, 2-Period, Open-label Crossover Study in Healthy Subjects to Determine the Effect of a Moderate CYP3A4 Inducer on the Pharmacokinetics of Omaveloxolone
Brief Title: An Open-label DDI Study of Omaveloxolone in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Celerion (Industry); Q2 Solutions (Industry); Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 408-C-2202
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adult Subjects
Keywords: omaveloxolone; DDI
MeSH Terms: interventions — omaveloxolone; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omaveloxolone only (Period 1), Then Omaveloxolone and efavirenz (Period 2) (Experimental): Period 1 (Day 1 - 15): Omaveloxolone Capsules, 150 mg, administered orally in a single dose on Day 1 Period 2 (Day 15 - 43): Efavirenz Tablet, 600 mg, administered orally once daily from Day 15 - Day 42 and Omaveloxolone Capsules, 150 mg, administered orally in a single dose on Day 29
  Interventions: Drug: Omaveloxolone; Drug: Efavirenz

INTERVENTIONS:
Drug: Omaveloxolone — Omaveloxolone Capsules, 150 mg, administered orally
  Other Names: RTA 408
Drug: Efavirenz — Efavirenz Tablet, 600 mg, administered orally once daily

SUMMARY:
This is an open-label, single-sequence, 2-period crossover study in healthy subjects.

In this study, 20 subjects will be enrolled to allow at least 16 evaluable subjects.

Subjects will receive a single oral dose of 150 mg omaveloxolone (3 × 50 mg capsules) on Day 1 (Period 1) and on Day 29 (Period 2), and 600 mg efavirenz once a day from Days 15 through 42 (Period 2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and/or females, 18 to 55 years of age (inclusive) at the time of screening.
* BMI at screening between 18.0 and 32.0 kg/m2 (inclusive)
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any major system disorder, as determined by the investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
* Use of any prescription medication before the first study drug administration (within 14 days before initial study drug administration or within 5 half-lives of the prescription medication, whichever is longer), and until after the last protocol-specified blood sample is prohibited, other than use of hormonal contraception.
* Clinically significant abnormal 12 lead ECGs
* Personal history of unexplained syncopal events, or family history of long QT syndrome or sudden unexplained death in a young person.
* Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines.
* History of drug or alcohol abuse in the last 6 months
* Positive hepatitis panel and/or positive human immunodeficiency virus test.
* Presence of hypotension (diastolic blood pressure ≤50 mmHg, systolic blood pressure ≤90 mmHg) or hypertension (diastolic blood pressure ≥ 140 mmHg, systolic blood pressure ≥ 90 mmHg)
* Blood donation (excluding plasma donation) within 56 days prior to screening and plasma donation within 7 days before screening.
* Positive urine drug screen or positive alcohol breath test result or positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of omaveloxolone | 43 days
  Blood samples to assess omaveloxolone PK will be collected predose and at the specified time points over a 336-hour period following each omaveloxolone dose for the duration of the study.
Area under the plasma concentration-time curve from 0 to tlast (AUC0-tlas) of omaveloxolone | 43 days
  Blood samples to assess omaveloxolone PK will be collected predose and at the specified time points over a 336-hour period following each omaveloxolone dose for the duration of the study.
Area under the plasma concentration-time curve from 0 extrapolated to infinity (AUC0-∞) of omaveloxolone | 43 days
  Blood samples to assess omaveloxolone PK will be collected predose and at the specified time points over a 336-hour period following each omaveloxolone dose for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Valentine, DO, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/